CLINICAL TRIAL: NCT01599260
Title: Resistance Exercise in Rheumatic Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding ended.
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NA_00069415
Record Dates: First submitted 2012-05-07; First posted 2012-05-15 (Estimated); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: Rheumatoid Arthritis; Systemic Vasculitis
MeSH Terms: conditions — Arthritis, Rheumatoid; Systemic Vasculitis | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Resistance Exercise (Experimental): Subjects will participate in a 16 week long resistance exercise program which will consist of 2 30-minute individually supervised sessions per week.
  Interventions: Other: Resistance Exercise

INTERVENTIONS:
Other: Resistance Exercise — Two 30-minute individually supervised exercise sessions per week for 16-weeks

SUMMARY:
People with rheumatic disease often have decreased strength, muscle mass, and bone mineral density due to repeated bouts of inflammation, normal effects of aging, disuse, and inactivity. The medications used to quell the disease process, such as prednisone, can also have detrimental effects on body composition, strength, and functional capacity. The investigators propose to investigate the feasibility, safety, and effects of resistance exercise in older patients with rheumatoid arthritis (RA) and vasculitis. The unique resistance protocol the investigators propose involves performing movements in a slow and controlled fashion (i.e., no acceleration or use of momentum in the lifting and lowering of the resistance) to minimize force on the joints and connective tissues. This will be conducted in an individually-supervised environment with a new generation of exercise equipment that will accommodate their musculoskeletal capabilities and allow for reproducibility of the exercise protocol. The investigators intend to investigate the feasibility, safety, musculoskeletal, and psychological effects of this resistance exercise protocol in older patients with rheumatoid arthritis and vasculitis by testing their strength, body composition, functional ability, mood, and quality of life before and after this 16-week resistance exercise intervention.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of rheumatoid arthritis OR systemic vasculitis (defined as granulomatosis with polyangiitis, Churg-Strauss, microscopic polyangiitis, Anti-neutrophil cytoplasmic autoantibody (ANCA)-associated vasculitis, or giant cell arteritis)

Exclusion Criteria:

* Non-English speaking
* Pregnancy
* Absolute cardiac or pulmonary contraindication to exercise
* pacemaker

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2012-05 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Number of participants with rheumatoid arthritis flares during the study | up to 16 weeks
  Participants will be provided with questionnaires. They will be asked to report the number of arthritis flares since the last visit. Arthritis flares consist of pain and swelling of the joints. The total number of flares during the 16 week study will be reported.
Number of participants with reported physical injuries during the study | up to 16 weeks
  Participants will be provided with questionnaires. They will be asked to report the number of injuries associated with the last visit (e.g. strains, sprains, and pulled muscles). The total number of injuries during the 16 week study will be reported.

SECONDARY OUTCOMES:
Change in Body composition after 16 weeks of resistance exercise | 16 weeks
  To assess change in body composition associated with this resistance exercise protocol (after 16 weeks).
Change in Strength after 16 weeks of resistance exercise | 16 weeks
  We will test if strength increases before and after the exercise intervention
Change in Functional status after 16 weeks of resistance exercise | 16 weeks
  We will determine if functional status, as measured by the short physical performance battery, improves after 16 weeks
Change in inflammatory cytokine Interleukin-6 (IL6) after 16 weeks of resistance exercise | 16 weeks
  Participants will have blood drawn before and after 16 weeks of exercise to determine if changes have occurred in their inflammatory cytokine.
Change in inflammatory cytokine C-reactive protein (CRP) after 16 weeks of resistance exercise | 16 weeks
  Participants will have blood drawn before and after 16 weeks of exercise to determine if changes have occurred in their inflammatory cytokine.
Change in Erythrocyte Sedimentation Rate (ESR) after 16 weeks of resistance exercise | 16 weeks
  Participants will have blood drawn before and after 16 weeks of exercise to determine if changes have occurred in their ESR

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca L Manno, M.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview Medical Campus, Baltimore, Maryland, United States